CLINICAL TRIAL: NCT07089758
Title: A Pilot Feasibility Study for Cerebral Open Flow Microperfusion in Patients Undergoing Planned Neurosurgical Resection of Diseased Parenchyma.
Brief Title: A Study for Cerebral Open Flow Microperfusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Terry Burns, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 25-001538; R37CA276851 (NIH)
Record Dates: First submitted 2025-07-25; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study Group (Experimental): Patients undergoing a planned neurosurgical resection of diseased brain parenchyma.
  Interventions: Device: Cerebral open flow microperfusion

INTERVENTIONS:
Device: Cerebral open flow microperfusion — Patients will undergo intra-operative microperfusion using Joanneum Research's cerebral open flow microperfusion (OFM) catheters, push and pull tubing, and MPP102-II pump. This process utilizes a probe (catheter) inserted into the parenchyma to collect analytes of any size and polarity from the microenvironment. The microperfusion pump peristaltically pushes and pulls perfusate with no net fluid-exchange when the pump heads are set at equal flow rates. As perfusate enters the tip of the microperfusion catheter, analytes are exchanged based on a gradient between the interstitial fluid and the perfusate. The sample is then recovered via the "pull" portion of the peristaltatic microperfusion pump, enabling constant sampling volumes and preventing loss of the perfusate into the tissue.
  The duration is 60-80 minutes (dependent on the speed of progress resecting portions of the tumor without catheters)
  Other Names: Joanneum Research cerebral open flow microperfusion

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of intra-operative microperfusion during a planned neurosurgical resection of diseased brain parenchyma, including either an epileptic focus requiring temporal lobectomy or a glioma. Devices used for microperfusion are Joanneum Research cerebral open flow microperfusion (OFM) catheters, push and pull tubing, and MPP102-II pump.

ELIGIBILITY:
Inclusion Criteria

* ECOG performance status (PS) 0, 1 or 2.
* Clinical and radiographic evidence diagnosis of glioma, or a prior diagnosis of glioma (suspected WHO grade II-IV), OR clinical evidence of epileptic foci requiring a temporal lobectomy.
* Clinical indication for resection as part of routine clinical care, with plan for this to be performed at Mayo Clinic (Rochester, MN).
* Able and willing to provide informed consent either signed by themselves or a legally authorized representative.

Exclusion Criteria

* Vulnerable populations: pregnant women, prisoners or the mentally handicapped.
* Patients who are not appropriate candidates for surgery due to current or past medical history or uncontrolled concurrent illness.
* Patients whom the surgeon deems to be at increased risk of adverse effects from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 year
  Number of patients who develop persistent adverse events deemed related (possibly, probably, definitely) to the insertion or use of microperfusate catheters. Adverse events will be measured by CTCAE 5.0.
Sample collection | 1 year
  Number of patients for whom at least 1 specimen containing > 10 μL microperfusate is successfully collected from 2 or more locations.

CONTACTS AND LOCATIONS:
Overall Officials: Terence Burns, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials